CLINICAL TRIAL: NCT07201051
Title: A Phase 2 Randomized, Double-blind, Placebo-controlled Study to Investigate Efficacy, Safety, Immunogenicity, and Pharmacokinetics, of GSK3862995B in Participants With Bronchiectasis
Brief Title: A Study to Assess the Effectiveness and Safety of GSK3862995B in Adults With Bronchiectasis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 223977; 2025-522892-27-00 (EU CTIS Number)
Record Dates: First submitted 2025-09-23; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Bronchiectasis
Keywords: GSK3862995B; Bronchiectasis; Efficacy; Safety; Immunogenicity; Pharmacokinetics
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: This is double-blind placebo-controlled study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- GSK3862995B Dose Level 1 (Experimental): Participants will receive GSK3862995B Dose level 1.
  Interventions: Drug: GSK3862995B
- GSK3862995B Dose Level 2 (Experimental): Participants will receive GSK3862995B Dose level 2.
  Interventions: Drug: GSK3862995B
- Placebo (Placebo Comparator): Participants will receive matching placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK3862995B — Participants will be administered with dose level 1 of GSK3862995B.
  Arms: GSK3862995B Dose Level 1; GSK3862995B Dose Level 2
Drug: Placebo — Participants will be administered with matching placebo.
  Arms: Placebo

SUMMARY:
This study is designed to find out how effective and safe a new drug, GSK3862995B, is for adult participants with bronchiectasis, a chronic lung disease. The study will also test how the body processes the drug and to check for any immune reactions. Participants will be divided into groups randomly to receive either one of two different doses of the study drug or a placebo. The main goal of the study is to see how well the drug works compared to the placebo in helping those with bronchiectasis.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 18-35 kilograms per square meters (kg/m^2)
* Clinical history consistent with bronchiectasis (cough, chronic sputum production, and/or recurrent respiratory infections) that is confirmed on chest computed tomography (CT)
* Meet one of the two criteria:

  * In the 12 months prior to screening, have had 2 or more documented pulmonary exacerbations that required a new antibiotic prescription by a physician or 1 pulmonary exacerbation that required hospitalization; or
  * In the 12 months prior to screening, have had 0 or 1 pulmonary exacerbation and a QOL-B RSS of less than (<)50 at screening
* Current sputum producers
* Post-bronchodilator FEV1 greater than or equal to (>=) 30 percent (%) or greater of predicted normal value
* Non-smokers or former cigarette smokers
* Males and females of childbearing and non-childbearing potential
* A female participant is eligible to participate if she is not pregnant or breastfeeding
* Is a Woman of non-childbearing potential (WONCBP) or is a Woman of childbearing potential (WOCBP) and using a contraceptive method that is highly effective, with a failure rate of <1
* A WOCBP must have a negative highly sensitive serum pregnancy test within 28 days before the first dose of study intervention
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the Informed consent form (ICF) and in this protocol

Exclusion Criteria:

* Participants with a primary diagnosis of asthma or Chronic Obstructive Pulmonary Disorder (COPD) as judged by the investigator
* Bronchiectasis due to cystic fibrosis, alpha-1-antitrypsin deficiency, common variable immunodeficiency, hypogammaglobinemia, or traction bronchiectasis due to fibrotic lung disease
* Active non-tuberculosis mycobacterial (NTM) lung infection on treatment or meeting ATS/Infectious Diseases Society of America (IDSA) criteria for active lung infection
* Active tuberculosis, untreated latent Tuberculosis (TB), invasive fungal lung infections or allergic bronchopulmonary aspergillosis needing treatment
* Participant uses long-term oxygen therapy for more than 12 hours per day
* Participants with an acute lower respiratory tract pulmonary infection needing treatment or pulmonary exacerbation within 4 weeks of the screening visit.
* Participant has a past or current medical condition(s) or disease(s) that is/are not well controlled and, which in the judgment of the Investigator, may affect participant safety or affect study endpoints
* Participants with an unstable cardiac disease, myocardial infarction, Cerebrovascular Accident (CVA), stroke or New York Heart Association Class III or IV heart failure within 12 months prior to screening
* Participants with clinically significant abnormal Electrocardiogram (ECG) at screening which in the judgment of the Investigator, may affect participant safety or affect study endpoints
* Significant allergies to humanized monoclonal antibodies
* Participants with a history of lymphoma, leukemia, or any malignancy within the past 5 years, except for basal cell or squamous epithelial carcinomas of the skin that have been resected for cure with no evidence of recurrence or metastatic disease for 1-year
* A known or suspected immunodeficiency that has led to opportunistic infections, recurrent invasive infections, or prolonged infections that suggest an underlying immunocompromised state by the judgement of the investigator. Positive HIV antibody test
* Alanine aminotransferase (ALT) >2x Upper limit of normal (ULN)
* Total bilirubin >1.5xULN; Participants with Gilbert's syndrome can be included with total bilirubin >1.5xULN as long as direct bilirubin is less than or equal to (<=)1.5xULN
* Current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* Presence of hepatitis B surface antigen (Hepatitis B surface antigen [HBsAg]) and/or hepatitis B core antibody (Hepatitis B core antibody [HBcAb]) at screening or within 3 months prior to first dose of study intervention
* Positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study intervention
* Positive hepatitis C Hepatitis B core antibody (RNA) test result at screening or within 3 months prior to first dose of study intervention
* Corrected QT interval (QTc) >450 milliseconds (msec) at screening visit based on the average of triplicate ECGs The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-09-26 (Estimated); Primary Completion 2027-03-15 (Estimated); Study Completion 2027-11-08 (Estimated)

PRIMARY OUTCOMES:
Annualized rate of Exacerbations for GSK3862995B Dose Level 1 Following Repeat Doses Compared with Placebo | Up to Week 48
  Annualized rate of exacerbations for GSK3862995B dose 1 following repeat doses compared with placebo in participants with bronchiectasis will be evaluated.

SECONDARY OUTCOMES:
Annualized rate of Exacerbations for GSK3862995B Dose Level 2 Following Repeat Doses Compared with Placebo | Up to Week 48
  Annualized rate of exacerbations for GSK3862995B dose 2 following repeat doses compared with placebo in participants with bronchiectasis will be evaluated.
Time to first Exacerbation for GSK3862995B Dose Level 2 and Dose Level 1 Compared to Placebo | Up to Week 48
Annualized Rate of Severe Exacerbations for GSK3862995B Dose Level 1 and Dose Level 2 Compared to Placebo | Up to Week 48
  Annualized rate of exacerbations for GSK3862995B dose 1 and dose 2 compared to placebo will be evaluated.
Change from Baseline in Quality-of-life bronchiectasis respiratory symptom scale score (QOL-B RSS) | Baseline up to Week 48
  QOL-B questionnaire is a self-administered, patient-reported outcome measure assessing symptoms, functioning and health-related quality of life for participants with bronchiectasis. The scale contains 37- items with 8 scales (respiratory symptoms, physical, role, emotional and social functioning). Scores range from 0 to 100, with higher scores indicating a better quality of life.
Change from Baseline in St. George's Respiratory Questionnaire (SGRQ) | Baseline up to Week 48
  The SGRQ is a 50-item patient reported outcome measure designed to measure health impairment by addressing the frequency of respiratory symptoms and the participant's current state. The SGRQ allows for the calculation of a total score as well as 3 subscale scores (symptoms, activity, and impact on daily life). Higher scores indicate greater impairment of health.
Change from Baseline in Post-bronchodilator Forced expiratory volume in one second (FEV1) value | Baseline up to Week 48
  Change from baseline in post-bronchodilator FEV1 value will be reported.
Number of Participants with Serious Adverse Events (SAE) | From screening (Day -1) up to Week 72
  Number of participants with SAEs will be reported.
Number of Participants with of Adverse Events (AE) | From randomization (Day 1) to Week 72
  Number of Participants with AEs will be reported.
Number of Participants with Clinically Significant Changes from Baseline in Clinical Laboratory Parameters | Up to Week 72
  Number of participants with clinically significant changes in laboratory data (hematology, chemistry, and urinalysis) will be reported.
Number of Participants with Clinically Significant Changes from Baseline in Vital Signs | Up to Week 72
  Number of participants with clinically significant changes from baseline in vital signs will be reported.
Number of Participants with Clinically Significant Changes from Baseline in 12-lead Electrocardiogram (ECG) | Up to Week 72
  Number of participants with clinically significant changes from baseline in 12-lead electrocardiogram will be reported.
Serum Concentration of GSK3862995B | Week 1 up to Week 48
  Serum concentration of GSK3862995B following repeated dose level 1 and dose level 2 will be reported.
Number of Participants with Anti-drug Antibodies (ADAs) Against GSK3862995B | Up to Week 72
  Number of participants with ADA against GSK3862995B following repeated dose level 1 and dose level 2 will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
Study Sponsor will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or asset(s) with development terminated across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf